CLINICAL TRIAL: NCT06303817
Title: Double Knots Versus Triple Knots Facia Closure Method During Cesarean Section; is There a Difference in Pain Sensation or Cosmetic Satisfaction?
Brief Title: Double Knots Versus Triple Knots Facia Closure Method; is There a Difference in Pain Sensation or Cosmetic Satisfaction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fikriye Isil Adıguzel, Medical Doctor, Adana City Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1812
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section; Pain; Cosmetics Sensitivity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double knots group (Other): The edge of the fascia was determined with a Kocher clamp. The fascia was closed starting from the opposite side with a synthetic absorbable multifilament suture in a continuous fashion up to the Kocher clamp and tied the knots with the same single suture.
  Interventions: Other: Double knots facia closure method during cesarean section
- Triple knots group (Other): The edge of the fascia was fixed with the same suture material instead of the Kocher clamp, and the fascia was closed similarly, starting from the opposite corner via the second loop. Then the loops from the first suture were tied to the second suture.
  Interventions: Other: Triple knots facia closure method during cesarean section

INTERVENTIONS:
Other: Double knots facia closure method during cesarean section — In Group I (double knots group), the edge of the fascia was identified with a Kocher clamp. A synthetic absorbable multifilament suture was used to close the fascia in a continuous fashion, starting from the opposite side up to the Kocher clamp. The knots were tied with the same single suture. I
  Arms: Double knots group
Other: Triple knots facia closure method during cesarean section — n Group II (triple knots group), the edge of the fascia was fixed with the same suture material instead of the Kocher clamp. The fascia was closed similarly, starting from the opposite corner via the second loop. The loops from the first suture were tied to the second suture.
  Arms: Triple knots group

SUMMARY:
The study included women who were scheduled for an elective or had an emergency cesarean section. Age, body mass index (BMI), obstetric history, education status, smoking status and C-section indications of the patients were recorded. Patients with a previous suprapubic scar, medical conditions affecting wound healing (such as diabetes or chronic corticosteroid use), those needing a vertical incision (e.g., placenta previa), individuals with postoperative wound infection or under 18 years old were excluded. Data were collected in standardized data form by a research assistant. Pre- and post-surgery treatments and/or interventions were standardized. All patients received antimicrobial prophylaxis with cefazolin before the operation. The abdomen was entered via a transverse suprapubic skin incision and the surgical steps up to the point of facia closure were accomplished in a standard fashion. Technical differences such as blunt and sharp dissection, uterus exteriorization vs in situ, or parietal peritoneum closure were left to the surgeon's discretion. The procedures for facia closure are as follows; in Group I (Double knots group), the edge of the fascia was determined with a Kocher clamp. The fascia was closed starting from the opposite side with a synthetic absorbable multifilament suture in a continuous fashion up to the Kocher clamp and tied the knots with the same single suture (Figure 2; a-b). In Group II (Triple knots group), the edge of the fascia was fixed with the same suture material instead of the Kocher clamp, and the fascia was closed similarly, starting from the opposite corner via the second loop. Then the loops from the first suture were tied to the second suture (Figure 2; c-d). After the incision was irrigated with sterile saline solution, the subcutaneous space was closed if the thickness was 2 cm or more. Skin closure was accomplished with a subcuticular technique using a non-absorbable monofilament suture, which was removed on the 10th day postoperatively. A closed subcutaneous suction drain was not used in any of the patients. Postoperative pain at and around the incision line was measured on the 1st, and 10th days postoperatively on the NRS (Numeric Rating Scale), with "0" being "no pain" and "10" being "the worst pain imaginable." The 1st measurements were made face-to-face, and the 10th-day evaluation was made via telephone interviews by the same research assistant.

DETAILED DESCRIPTION:
This prospective randomized control trial was conducted in a single tertiary center between March 2022 and July 2022. The institutional ethics committee approved the study (Decision Number: 1812/2022), and all participants provided written informed consent. When determining the sample size, since there was no literature information, type I error was taken as 1%, the power of the test was taken as 90%, and the effect size between group I and group 2 was taken as 0.50 (moderated), a minimum of 106 people in each group and 212 people in total were included in the study (5). The study included women who were scheduled for an elective or had an emergency cesarean section. Age, body mass index (BMI), obstetric history, education status, smoking status and C-section indications of the patients were recorded. Patients with a previous suprapubic scar, medical conditions affecting wound healing (such as diabetes or chronic corticosteroid use), those needing a vertical incision (e.g., placenta previa), individuals with postoperative wound infection or under 18 years old were excluded. Data were collected in standardized data form by a research assistant.

The surgeons who participated in the study were obstetricians or senior residents and performed surgeries on patients in all groups and were not blinded because of the nature of the operative procedure. A block randomization with a block size of 4-6 and a ratio of 1:1 was applied. Sealed opaque envelopes were used for allocation concealment. Scrub nurses opened the envelopes in the operative room just before the skin incision.

Pre- and post-surgery treatments and/or interventions were standardized. All patients received antimicrobial prophylaxis with cefazolin before the operation. The abdomen was entered via a transverse suprapubic skin incision and the surgical steps up to the point of facia closure were accomplished in a standard fashion. Technical differences such as blunt and sharp dissection, uterus exteriorization vs in situ, or parietal peritoneum closure were left to the surgeon's discretion. The procedures for facia closure are as follows; in Group I (Double knots group), the edge of the fascia was determined with a Kocher clamp. The fascia was closed starting from the opposite side with a synthetic absorbable multifilament suture in a continuous fashion up to the Kocher clamp and tied the knots with the same single suture (Figure 2; a-b). In Group II (Triple knots group), the edge of the fascia was fixed with the same suture material instead of the Kocher clamp, and the fascia was closed similarly, starting from the opposite corner via the second loop. Then the loops from the first suture were tied to the second suture (Figure 2; c-d). After the incision was irrigated with sterile saline solution, the subcutaneous space was closed if the thickness was 2 cm or more. Skin closure was accomplished with a subcuticular technique using a non-absorbable monofilament suture, which was removed on the 10th day postoperatively. A closed subcutaneous suction drain was not used in any of the patients.

Postoperative pain at and around the incision line was measured on the 1st, and 10th days postoperatively on the NRS (Numeric Rating Scale), with "0" being "no pain" and "10" being "the worst pain imaginable." The 1st measurements were made face-to-face, and the 10th-day evaluation was made via telephone interviews by the same research assistant. In our clinic, we apply paracetamol 500 mg IV and diclofenac sodium intramuscularly (IM) to our patients postoperatively for pain management. Accumulative dosages of requested NSAİ and paracetamol during the hospital stay were also recorded. Patient satisfaction with the aesthetic results was assessed using a 10-point scale ranging from 1 (very unsatisfied) to 10 (very satisfied) at the 1st and 3rd months postoperatively. While scoring, patients were asked to score their scars by being reminded of parameters such as color, stiffness, thickness and irregularity. All patients were blinded to which technique was used for facial closure.

Statistical analysis Data were analyzed with IBM SPSS V23 (IBM Corp., Armonk, NY, USA). The normality assumptions were examined with the Kolmogorov-Smirnov test. Mann-Whitney U test was used to compare non-normally distributed data in pairs. Wilcoxon test was used to compare non-normally distributed data within groups according to two dependent times. Pearson chi-square, Yates correction, and Fisher's Exact Test were used to examine categorical variables according to groups. Data are expressed as mean (standard deviation, SD) or median (minimum-maximum), as appropriate. P <.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* women who were scheduled for an elective or had an emergency cesarean section

Exclusion Criteria:

* A previous suprapubic scar
* Medical conditions affecting wound healing (such as diabetes or chronic corticosteroid use)
* Those needing a vertical incision (e.g., placenta previa)
* Individuals with postoperative wound infection
* Under 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on NRS (Numeric Rating Scale) at 10 days | 1. and 10. day
  Postoperative pain at and around the incision line was measured on the 1st, and 10th days postoperatively on the NRS (Numeric Rating Scale), with "0" being "no pain" and "10" being "the worst pain imaginable."
Change from baseline in aesthetic results at 3 months | 1. day and 3. months
  . Patient satisfaction with the aesthetic results was assessed using a 10-point scale ranging from 1 (very unsatisfied) to 10 (very satisfied) at the 1st and 3rd months postoperatively. While scoring, patients were asked to score their scars by being reminded of parameters such as color, stiffness, thickness and irregularity. All patients were blinded to which technique was used for facial closure.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Baş, M.D., Study Director — Adana City Training and Research Hospital
Locations (1):
- Adana Şehir Eğitim ve Araştırma Hastanesi, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No